CLINICAL TRIAL: NCT00854542
Title: Effectiveness of Telepsychiatry-based Culturally Sensitive Collaborative Treatment of Depressed Chinese Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Albert Yeung, Albert Yeung, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008P001437
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Depression
Keywords: Telepsychiatry; Culturally Sensitive Collaborative Treatment; Chinese Americans; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TCSCT (Active Comparator)
  Interventions: Behavioral: Telepsychiatry-based Culturally Sensitive Collaborative Treatment
- Usual Care (Placebo Comparator)
  Interventions: Behavioral: Telepsychiatry-based Culturally Sensitive Collaborative Treatment

INTERVENTIONS:
Behavioral: Telepsychiatry-based Culturally Sensitive Collaborative Treatment — T-CSCT: Patients in Group A will receive T-CSCT, which consists of Telepsychiatry-based Culturally Sensitive Psychiatry Assessment using the Engagement Interview Protocol (EIP) plus Care Management.

SUMMARY:
Hypothesis 1. Telepsychiatry consultations will be acceptable and well-received by depressed Chinese Americans and by their primary care clinicians.

Hypothesis 2. Depressed Chinese Americans in remote primary care clinics receiving T-CSCT will have improved outcomes compared to patients who receive Usual Care by primary care physicians.

DETAILED DESCRIPTION:
Telepsychiatry-based CSCT (T-CSCT):

Live and interactive Telepsychiatry (using videoconferencing) brings tremendous opportunities to clinical care, education, research, and administration. In the U.S. to date, telepsychiatry has been implemented in rural areas where people lack access to psychiatrists (Baer et al, 1997), in the Prison System with service users constrained from traveling (Brecht et al., 1996), in rural native American resettlement areas (Shore & Spero, 2005), and in Alaska where residents are faced with both distance and a shortage of mental health professionals. In this proposed study, we plan to investigate the effectiveness of telepsychiatry-based CSCT (T-CSCT) to provide culturally sensitive collaborative management of MDD to monolingual Chinese Americans. For this group of patients, telepsychiatry consultation could be a necessity both in urban as well as rural primary care clinics that are not staffed with bilingual psychiatrists. T-CSCT plans to utilize the advanced telemedicine technology in major academic centers to connect the scarce resource of bilingual and bicultural mental health professionals to underserved Chinese Americans to improve their access to treatment of MDD.

T-CSCT will explore the usefulness and effectiveness of recognizing MDD subjects through consumer-initiated depression self-screening using the validated CB-PHQ-9, which will be made available in community newspapers, journals, and on the internet. To facilitate care management for Chinese Americans, a Depression Toolkit for Chinese Americans will be developed, which will include information on the nature and treatment of MDD, the CB-PHQ-9 for depression self-screening, a bilingual instrument to monitor progress of depressive symptoms, strategies for patients to negotiate with health professionals for individually tailored treatment for depression, and answers to frequently asked questions (FAQs) by Asian American immigrants on MDD and its treatment. If shown to be effective, the T-CSCT can be the prototype of a telemedicine-based Multiracial Mental Health Resource Center to provide services to other minority populations to reduce disparities in mental health treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with Chinese ethnicity, defined as people who self-identify as being Chinese based upon having either one or both parents being ethnic Chinese.
2. Monolingual Chinese American immigrants, defined as people who require or prefer to be interviewed in Chinese (including Cantonese, Taiwanese, Mandarin, and Toisanese dialects).
3. Men or women age 18 or older, who live in the greater Boston area.
4. Individuals who are competent to consent and have completed a written consent form.
5. Individuals who have a PCP.
6. Patients who screen positive for MDD, current according to the fourth version of the Diagnostic and Statistical Manual for Mental Disorders (DSM-IV) as diagnosed by the Mini International Neuropsychiatric Interview (MINI; Sheehan et al, 1998)
7. Individuals who are willing to receive phone interviews for monitoring of symptoms and for additional support (care management) if available.

Exclusion Criteria:

1. Patients with serious suicidal risk.
2. Patients with unstable medical illnesses requiring imminent hospitalization or rendering patients unsuitable for clinical interview.

d. Patients with comorbid severe mental disorders including:

1. Organic mental disorders.
2. Alcohol or substance abuse disorders active within the last year.
3. Schizophrenia.
4. Delusional disorder.
5. Psychotic disorders not elsewhere classified.
6. Bipolar disorder. e. Patients with history of treatment by a psychiatrist in the past 4 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2009-01; Primary Completion 2014-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | Screen, Week 9, 17, 24

SECONDARY OUTCOMES:
Clinical Global Impressions (Severity of Depression and Global Improvement) | Screen, Week 9, 17, 24

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yeung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- South Cove Community Health Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Chen JA, Shapero BG, Trinh NT, Chang TE, Parkin S, Alpert JE, Fava M, Yeung AS. Association Between Stigma and Depression Outcomes Among Chinese Immigrants in a Primary Care Setting. J Clin Psychiatry. 2016 Oct;77(10):e1287-e1292. doi: 10.4088/JCP.15m10225. PMID 27631145
- [Derived] Yeung A, Martinson MA, Baer L, Chen J, Clain A, Williams A, Chang TE, Trinh NH, Alpert JE, Fava M. The Effectiveness of Telepsychiatry-Based Culturally Sensitive Collaborative Treatment for Depressed Chinese American Immigrants: A Randomized Controlled Trial. J Clin Psychiatry. 2016 Aug;77(8):e996-e1002. doi: 10.4088/JCP.15m09952. PMID 27561153
- [Derived] Yeung A, Hails K, Chang T, Trinh NH, Fava M. A study of the effectiveness of telepsychiatry-based culturally sensitive collaborative treatment of depressed Chinese Americans. BMC Psychiatry. 2011 Sep 26;11:154. doi: 10.1186/1471-244X-11-154. PMID 21943315